CLINICAL TRIAL: NCT00199355
Title: Placebo-Controlled , Double-Blind , Exploratory Study of KW-6002(Istradefylline) in the Treatment of Parkinson's Disease. [Adjunctive Therapy to Levodopa]
Brief Title: A Study of Istradefylline (KW-6002) for the Treatment of Parkinson's Disease in Patients Taking Levodopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-0406
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
To establish the efficacy of 20 mg/day and 40 mg/day doses of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa.

DETAILED DESCRIPTION:
To establish the efficacy of 20 mg/d and 40mg/d doses of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa. Patients who meet entry criteria will be randomized in a 1:1:1 ratio to double blind treatment with oral doses of 20 or 40mg/d istradefylline or matching placebo. Patients will be treated for 12 weeks and will have interim visits and end of treatment visit to assess the efficacy and safety of istradefylline.

ELIGIBILITY:
Inclusion Criteria:

1. UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD.
2. PD stages 2-4 in the OFF state for Modified Hoehn and Yahr Scale.
3. On levodopa/DCI for at least one year, stable dose in past 4 weeks.
4. Currently take at least three doses of levodopa/DCI per day.
5. Predictable end of dose wearing off.
6. Able to satisfactorily complete Hauser version of a Parkinson's diary.
7. Have an average of 120 minutes of OFF time on two 24 hour diaries.
8. On a stable regimen of medications being administered within normal therapeutic limits for Parkinson's disease for at least four weeks before randomization.
9. Be at least 30 years of age.

Exclusion Criteria:

1. Neurosurgical treatment for PD.
2. History of psychosis.
3. Diagnosis of atypical Parkinsonism or secondary Parkinsonism variant.
4. Diagnosis of cancer within 5 years.
5. Diagnosis of clinically significant illness of any organ system.
6. Mini-mental status examination score of 25 or less.
7. Taking any excluded medications.
8. History of drug or alcohol abuse or dependence within the past two years.
9. History of seizures or neurological malignant syndrome.
10. Clinical depression.
11. Pregnant or lactating females.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To establish the efficacy of 20 mg/d and 40mg/d doses of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa/DCI.

SECONDARY OUTCOMES:
To evaluate the efficacy of 20 mg/d and 40mg/d dose of istradefylline for reducing the total hours of OFF time.
To evaluate the change in percentage of ON time (without dyskinesia, with dyskinesia, with non-troublesome dyskinesia, and with troublesome dyskinesia).
To evaluate the change in Unified Parkinson's Disease Rating Scale (UPDRS).
To evaluate change in the Clinical Global Impression - Improvement scale (CGI-I).
To evaluate change in the Clinical Global Impression - Severity of Illness scale (CGI-S).
To evaluate the safety of 20 mg/d and 40mg/d doses of istradefylline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan